CLINICAL TRIAL: NCT04847752
Title: A Prospective Observational Cohort Study of Predictive Factors Related to Prognosis of In-hosiptal Patients With Ischemic Stroke Due to Large-artery Atherosclerosis
Brief Title: Study of Predictive Factors Related to Prognosis of Patients With Ischemic Stroke Due to Large-artery Atherosclerosis
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Daishi Tian, Prof., Tongji Hospital
Other Study IDs: TJID-20210404TDS
Record Dates: First submitted 2021-04-12; First posted 2021-04-19 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Ischemic Stroke; Large-Artery Atherosclerosis (Embolus/Thrombosis)
MeSH Terms: conditions — Ischemic Stroke; Embolism; Thrombosis | interventions — Endarterectomy, Carotid; Aspirin; Clopidogrel; Anticoagulants; Warfarin; Rivaroxaban; Dabigatran; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atorvastatin; Rosuvastatin Calcium; evolocumab; alirocumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — carotid plaque fixed tissues and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: carotid artery stenting — common treatments for carotid artery stenosis
  Other Names: CAS
Procedure: carotid endarterectomy — common treatments for carotid artery stenosis
  Other Names: CEA
Drug: Aspirin — the dosage and duration
  Other Names: ASP
Drug: Clopidogrel — the dosage and duration
  Other Names: plavix
Drug: Anticoagulant — the dosage and duration
  Other Names: warfarin; rivaroxaban; dabigatran; any other anticoagulant therapy
Drug: Statin — the dosage and duration
  Other Names: atorvastatin; rosuvastatin; any other statin drugs
Drug: PCSK9 inhibitor — the dosage and duration
  Other Names: Evolocumab; Alirocumab; any other PCSK9 inhibitors

SUMMARY:
This is a single-center prospective cohort study of predictive factors related to prognosis of ischemic stroke due to large-artery atherosclerosis.

From March 1, 2021 to December 31, 2026, 1000 patients with ischemic stroke due to large-artery atherosclerosis who are admitted to the Department of Neurology or Neurosurgery, Tongji Hospital are going to be recruited. Detailed clinical data in emergency room and in-hospital will be obtained from the medical record reviews, and the National Institutes of Health Stroke Scale (NIHSS) and Modified Rankin Scale (mRS) score will be done by certified neurologists to assess the severity of the disease in acute stage and treatment outcome during the follow-up. All cases will undergo routine blood tests, brain magnetic resonance imaging (MRI) and cerebral vascular examination, such as TCD, CTA, HRMR or DSA. The investigators will analyze the in-hospital factors that could predict the outcome to provide more evidence-based suggestions in the treatment and prognosis of atherosclerotic ischemic cerebrovascular disease.

DETAILED DESCRIPTION:
The detaited information about this trial is described below

1. Quality assurance: The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
2. Data check: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data.
3. Source data verification: Medical records, electronic case report forms, and imaging would be processed by certified neurologists.
4. Data included:

   4.1 Baseline Variables: NIHSS and mRS scores before ischemic stroke 4.2 In-hospital Variables: 4.2.1 Main symptoms（1=facial paralysis 2=limb weakness 3=limb numbness 4=facial numbness 5=lalopathy 6=ataxia 7=dysphagia 8=bulbar paralysis 9=dizziness 10=nausea and vomit 11=vision disorder 12=confusion 13=headache 14=unconsciousness 15=others） NIHSS and mRS scores after admission 4.2.2 Brain CT and ASPECT scores 4.2.3 DWI 4.2.4 CTA, MRA, DSA, carotid artery ultrasound andTCD to evaluate the stenosis degree of large vessels 4.2.5 HRMR to evaluate the changes of the plaque of intracranial stenosis 4.2.6 Blood routine tests 4.2.7 HbALc and FBG 4.2.8 LDL HDL ApoA1 and ApoB 4.2.9 Cardiac TnI and NT-proBNP 4.2.10 Proteomic analysis of fresh plasma 4.2.11 Histopathological tissues and transcriptomics of CEA
5. Standard Operating Procedures 5.1 Patient recruitment: From March 1, 2021 to December 31, 2026, 1000 patients with ischemic stroke due to large-artery atherosclerosis who are admitted to the Department of Neurology and Neurosurgery, Tongji Hospital are going to be recruited 5.2 Data collection: Detailed clinical data in emergency room and in-hospital will be obtained from the medical record reviews, and the National Institutes of Health Stroke Scale (NIHSS) and Modified Rankin Scale (mRS) score will be done by certified neurologists to assess the severity of the disease in acute stage and clinical outcome during the follow-up. All cases would undergo routine blood tests, brain magnetic resonance imaging (MRI) and cerebral vascular examination, such as TCD, CTA, HRMR or DSA.

   5.3 Data management, The research data is reviewed by an Independent Research Panel.

   5.4 Data analysis: Biostatisticians from the Department of Neurology, Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology will conduct statistical analysis
6. Sample size assessment: About 1000 cases.
7. Plan for missing data: The number of lost cases will be treated as the deleted value and the lost rate will be indicated. Complete sample intentionality analysis and intent-to-treat (ITT) analysis would be performed on the end points. During the analysis, if there is a statistical difference in the results, the number of participants lost in the exposed group will be deleted, and the number of participants lost to in the non-exposed group will be added. If there is still a statistical difference in the results, the loss of follow-up will not have an impact on the analysis results of this group.
8. Statistical analysis: All statistical data would be analyzed by the SPSS Software 24.0 version. Continuous variables would be reported as median (range, minimum-maximum), which would be compared by Mann-Whitney test, and categorical data would be represented as percentages and frequencies, which would be compared by the two-tailed Fisher's exact test or one-way ANOVA. P<0.05 would be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke due to large-artery atherosclerosis has been proved by clinical symptoms and imaging examinations.
* Symptomatic superior arch stenosis >50%
* Asymptomatic superior arch stenosis was >70%
* written informed consent was obtained from patients or their surrogates before enrollment.

Exclusion Criteria:

* Brain CT or MRI showing cerebral hemorrhage (excluded ischemic stroke with hemorrhage transformation)
* With severe systemic disease, are expected to survive < 3 months
* Patients will not able to provide continuous follow-up information

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ischemic stroke due to large-artery atherosclerosis admission to Department of Neurology and Neurosurgery, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology from March 1, 2021 - December 31, 2026
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | 3-6 months after onset.
  Death during the follow-up in every single reason
Stroke of any kind | 3-6 months after onset.
  Brain CT or MRI scans will be used to measure whether there is any kind of stroke, including TIA, ischemic stroke, and hemorrhage

SECONDARY OUTCOMES:
Rehospitalization | 1 month to 24 months after onset.
  The rehospitalized times of any circumstances except for admission to hospital only for examination per year will be used to measure the situation
National Institute of Health stroke scale (NIHSS score) | 1 month to 24 months after onset.
  The minimum value is 0, and maximum value is 42, and higher scores mean a worse outcome.
modified Ranking score (mRS) | 1 month to 24 months after onset.
  The minimum value is 0, and maximum value is 6, and higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dai-Shi Tian, Dr., Study Chair — Tongji Hospital; Chuan Qin, Dr., Principal Investigator — Tongji Hospital; Jun Xiao, Dr., Principal Investigator — Tongji Hospital; Ke Shang, Dr., Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: starting 12 months after publication
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.